CLINICAL TRIAL: NCT07332715
Title: Predictive Value of the Combination of Uric Acid/Albumin Ratio and Lactate for Acute Kidney Injury, Hemodynamic Support Requirement, and Mortality in Patients With Sepsis
Brief Title: Predictive Value of the Uric Acid/Albumin Ratio and Lactate in Sepsis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assos.Prof., Istinye University
Other Study IDs: 330-2025
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Sepsis-Related Mortality; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional / Observational Study — This is a non-interventional, observational study. No diagnostic or therapeutic intervention will be applied beyond routine clinical care. Blood uric acid, albumin, and serum lactate levels measured as part of standard intensive care management will be recorded at admission, and lactate levels will be reassessed at 24 hours. Patients will be followed prospectively during their intensive care stay to evaluate the development of acute kidney injury, vasopressor requirement, and 28-day mortality.

SUMMARY:
Sepsis is a life-threatening condition characterized by organ dysfunction resulting from a dysregulated host response to infection and remains a leading cause of morbidity and mortality in intensive care units. Early identification of patients at high risk for adverse outcomes is essential for timely intervention and improved prognosis.

This prospective, single-center, non-interventional study aims to evaluate the predictive value of the combined use of the blood uric acid/albumin ratio (UAR) and serum lactate levels in patients aged 65 years and older who are admitted to the intensive care unit with a diagnosis of sepsis according to SEPSIS-3 criteria. Patients without acute kidney injury at admission and with at least 24 hours of intensive care follow-up will be included.

The primary outcome is the development of acute kidney injury within the first 7 days of ICU admission according to KDIGO criteria. Secondary outcomes include vasopressor requirement during ICU stay, changes in serum lactate levels over the first 24 hours, and 28-day mortality. The study seeks to determine whether the combination of UAR and lactate levels can serve as an easily accessible and clinically applicable biomarker to predict adverse outcomes and support prognostic assessment and treatment strategies in sepsis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older
* Diagnosis of sepsis according to SEPSIS-3 criteria
* Admission to the intensive care unit
* No acute kidney injury at admission according to KDIGO classification
* Measurement of serum uric acid, albumin, and lactate levels at ICU admission
* SOFA score calculated at ICU admission
* ICU follow-up of at least 24 hours

Exclusion Criteria:

* Age under 65 years
* Uncompensated or decompensated chronic liver disease (e.g., Child-Pugh class C)
* Chronic kidney disease stage 4 or 5 (eGFR <30 mL/min/1.73 m²)
* Presence of acute kidney injury at admission according to KDIGO criteria
* Active malignancy or receipt of active cancer treatment within the last 6 months
* Missing or incomplete clinical/laboratory data
* ICU follow-up less than 24 hours

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of critically ill adult patients aged 65 years and older who are admitted to a tertiary-level intensive care unit with a diagnosis of sepsis based on SEPSIS-3 criteria. All participants are required to have baseline measurements of serum uric acid, albumin, and lactate levels at the time of ICU admission and no evidence of acute kidney injury at presentation. The study focuses on evaluating the prognostic value of routinely available biochemical markers in predicting adverse clinical outcomes, including acute kidney injury, vasopressor requirement, and short-term mortality during intensive care follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Development of Acute Kidney Injury (AKI) | Within the first 7 days following intensive care unit admission
  Occurrence of acute kidney injury defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria in patients with sepsis admitted to the intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

REFERENCES:
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Barichello T, Generoso JS, Singer M, Dal-Pizzol F. Biomarkers for sepsis: more than just fever and leukocytosis-a narrative review. Crit Care. 2022 Jan 6;26(1):14. doi: 10.1186/s13054-021-03862-5. PMID 34991675